CLINICAL TRIAL: NCT06378060
Title: A Prospective, Multi-center, Single-arm Clinical Study to Evaluate the Safety and Efficacy of a Modified Allogeneic Hematopoietic Stem Cell Transplantation Regimen for Severe Aplastic Anemia
Brief Title: Clinical Study on Modified Allogeneic Hematopoietic Stem Cell Transplantation Regimen for Severe Aplastic Anemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hematology department of the 920th hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM04
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-03

CONDITIONS: Severe Aplastic Anemia
Keywords: Severe Aplastic Anemia; Modified transplantation system; Ruxolitinib; Melphalan
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Modified transplantation system

INTERVENTIONS:
Drug: Modified transplantation system — Conditioning regimen: fludarabine 30mg/m2×5~6d,cyclophosphamide 50mg/kg×2d, melphalan 100mg/m2×1d aGVHD prophylaxis: PTCY 25mg/kg×2d, ATG 4.5mg/kg total, MMF 15mg/kg +5d~+35d, Ruxolitinib 5mg bid -1d~+50d and 2.5mg bid +51d~+110d, CSA

SUMMARY:
The aim of this study was to evaluate the safety and efficacy of a modified allogeneic hematopoietic stem cell transplantation regimen for aplastic anemia.

DETAILED DESCRIPTION:
ObjectiveTo evaluate the safety and efficacy of a modified allogeneic hematopoietic stem cell transplantation regimen in aplastic anemia. Aplastic anemia (AA) is a group of myelo-hemopoietic failure syndromes caused by a variety of etiologies. If not intervened, the average expected survival time is less than half a year.Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is one of the possible cures for this disease. The success rate of treatment for this disease can be further improved under the previous regimen system. The survival rate reported in the literature is 60%-90%. We designed this study to improve the conditioning regimen and optimize the GHVD prevention measures to improve the transplant success rate and prolong patient survival, while minimizing the occurrence of GVHD and reducing the recurrence rate of the disease.30 patients with aplastic anemia were planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with benign or malignant hematological diseases such as leukemia, lymphoma, thalassemia, aplastic anemia, etc. diagnosed by NCCN guidelines, and requiring allogeneic hematopoietic stem cell transplantation as determined by the researchers;
2. Age 3-65 years old;
3. Weight 10Kg-100Kg;
4. Eastern Cooperative Oncology Group (ECOG) score ≤3;
5. No major organ injury (ECG ejection fraction >45%; bilirubin < 2 times the upper limit of normal value; AST and ALT < 3 times the upper limit of normal value; serum creatinine < 2 times the upper limit of normal value);
6. No severe infection;
7. Subjects voluntarily participated in this clinical trial and signed the informed consent.

Exclusion Criteria:

1. patients with nonhematologic diseases who are not eligible for transplantation or who do not wish to receive transplantation;
2. patients with an expected survival of less than 1 month;
3. patients with previous autologous or allogeneic hematopoietic stem cell transplantation;
4. pregnant patients;
5. patients with severe mental or neurological disorders that would affect the ability to provide informed consent and/or to report or observe adverse events;
6. other conditions that the investigator determines to be inappropriate for enrollment.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | [Time Frame: 2 years after allogeneic transplantation with improved conditioning regimen]
  2-year overall survival (OS) and graft-versus-host disease and relapse-free survival (GRFS) after transplantation
Acute graft-versus-host disease incidence | [Time Frame: 2 years after allogeneic transplantation with improved conditioning regimen]

SECONDARY OUTCOMES:
Transplantation-related motality | [Time Frame: 2 years after allogeneic transplantation with improved conditioning regimen]
Chronic graft-versus-host disease incidence | [Time Frame: 2 years after allogeneic transplantation with improved conditioning regimen]
incidence of Intensive fungal disease | [Time Frame: 2 years after allogeneic transplantation with improved conditioning regimen]
EB virus reactivation rate | [Time Frame: 2 years after allogeneic transplantation with improved conditioning regimen]
CMV reactivation rate | [Time Frame: 2 years after allogeneic transplantation with improved conditioning regimen]

CONTACTS AND LOCATIONS:
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No